CLINICAL TRIAL: NCT02228629
Title: Do CrocsRx Clogs Reduce Dynamic Plantar Pressure as Compared to Conventional House Shoes in Subjects With Diabetes?
Brief Title: Utility of CrocsRx Clog as a Diabetic House Shoe: a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Responsible Party: Principal Investigator, Jinsup Song, Director, Gait Study Center, Temple University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21391
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes
Keywords: Diabetes; Foot complications; plantar keratoma; plantar pressure
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Typical house shoe (Experimental): Subject's typical shoes worn in and around home
  Interventions: Device: CrocsRx Medical Silver cloud clogs

INTERVENTIONS:
Device: CrocsRx Medical Silver cloud clogs

SUMMARY:
Foot complications are a common and costly problem for subjects with diabetes. Although Medicare provides a pair of diabetic shoes yearly for subjects with diabetes, many do not wear their diabetic shoes in and around their house. Instead, subjects may wear shoes, such as flip flops or slippers, that provide little to no protection against injuries. While proper house shoe is important in the prevention of diabetic foot complications, this area has not received much attention. The purpose of this pilot study is to assess if CrocsRx Medical silver cloud clogs - a lightweight clog with protective toe box, cushioning soles, and easy to don and doff - offer reduced dynamic plantar pressure magnitude, as compared to conventional house shoes, for subjects with diabetes. A Repeated Measures ANOVA study design will be used to assess dynamic plantar pressure in 2 shod conditions for each subject with the order of shoes randomized.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 21 and 75 (inclusive)
* Documented type 1 or type 2 diabetes mellitus
* Demonstrated abnormal foot biomechanics by the presence of intractable plantar keratoma (IPK) beneath metatarsal heads or hallux
* Participants with and without signs of peripheral neuropathy (unable to perceive a 10 gram monofilament or vibration perception threshold (VPT > 25 Volts)
* Able to walk independently without the use of walking aids (cane, crutches, or walker)
* Able to speak and understand English
* Able to understand the information in the consent form and willing and able to sign the consent form

Exclusion Criteria:

* History of lower limb amputations (excluding toe amputations)
* Presence of cutaneous ulceration in the lower extremity
* History of or active Charcot neuroarthropathy of either foot
* Severe peripheral vascular disease (i.e. ischemic rest pain, 2-block claudication, or gangrene)
* End stage kidney disease requiring hemodialysis, stroke, or widespread malignant disease
* Pregnant or nursing
* Not willing or able to make the required follow-up visits
* Insufficient (corrected) vision to complete the questionnaire
* Unable to fit into available shoe sizes

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of peak pressure sub-metatarsal 2 and hallux in usual house shoes versus the CrocsRx clogs | At visit 1.
  In-shoe plantar pressures will be measured using novel pedar-X system on subjects with diabetes while walking in 2 shod conditions: (1) their usual house shoe and (2) the CrocsRx clogs.

CONTACTS AND LOCATIONS:
Locations (1):
- Gait Study Center at the Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania, United States